CLINICAL TRIAL: NCT04057729
Title: An Open-label, Randomized, Single-dose, Two-way Crossover Study to Evaluate the Effect of Food on the Pharmacokinetic Characteristics of IMP4297 Capsules in Healthy Subjects
Brief Title: IMP4297 Food Effect Trial in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Impact Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: IMP4297-103
Record Dates: First submitted 2019-07-29; First posted 2019-08-15 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Solid Tumor
MeSH Terms: interventions — senaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 （IMP4297 100mg, Fasted-Fed） (Experimental): Period 1: Fasted control → Period 2: Fed control
  Interventions: Drug: IMP4297
- Arm 2（IMP4297 100mg, Fed- Fasted） (Experimental): Period 1: Fed control → Period 2: Fasted control
  Interventions: Drug: IMP4297

INTERVENTIONS:
Drug: IMP4297 — 10mg/capsule.

SUMMARY:
A phase I, single-site, open-label, randomized, single-dose, two-way crossover study to evaluate the effect of food on the pharmacokinetic characteristics of IMP4297 capsules in China

DETAILED DESCRIPTION:
This food-effect study plans to enroll 16 (at least 12 to complete the study) subjects. Subjects will be randomly assigned to 1 of 2 dosing sequences (fasted or standard high-fat breakfast) at a 1:1 ratio generated from a computer. Each dosing sequence will consist of 2 cycles, with 1 dose in each cycle of the study and a washout period of at least 7 days between each dose. Study drug will be administered to subjects in the morning of each administration day of each cycle. PK, ECG, vital signs, physical examinations and laboratory tests will be performed as specified in the protocol. Tolerability and safety of the treatment will be evaluated by monitoring adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Must fully understand the purpose, nature, methods of the trial and possible adverse reactions and volunteer as a subject. Subjects have to sign informed consent themselves prior to any study-related procedures and ensure that any procedure would involve themselves in the study.
2. Chinese male subjects aged 18 to 55 years (inclusive) at screening.
3. Have body mass index (BMI) between 19.0 and 26.0 kg/m2 (inclusive), and body weight≥50.0 kg.
4. Detailed medical history, vital signs (blood pressure, pulse and body temperature), comprehensive physical examination, laboratory tests (blood routine, blood biochemistry and urine routine), 12-lead electrocardiogram (ECG) and other test results show no abnormality or without clinical significance if abnormal.
5. Have no plan of giving birth and be willing to use effective contraception; and have no plan to donate sperm during the study and 90 days after the last dose of the investigational drug. Non-drug contraception should be used during the trial voluntarily.
6. Be able to communicate well with the investigator, understand and comply with the requirements of the study.

Exclusion Criteria:

1. Have clinical abnormalities to be excluded, including but not limited to disorders of the nervous system, cardiovascular system, blood and lymphatic system, immune system, kidney, liver, gastrointestinal tract, respiratory system, metabolism, bone and other systemic diseases.
2. Have a history of allergic disease (including drug allergies, allergic reactions to two or more foods).
3. Have a history of dysphagia or any gastrointestinal disorder affecting drug absorption.
4. Have had surgery within 3 months prior to screening or have scheduled surgery during the study, and have had surgery which may affect the absorption, distribution, metabolism and excretion of drugs.
5. Inability to tolerate venipuncture, have fear of needles and have a history of hemophobia.
6. Have lactose intolerance (who have had diarrhea after drinking milk).
7. History of drug abuse within 6 months prior to screening or a positive result on urine drug screen (baseline period).
8. History of using narcotic drugs within 3 months prior to screening.
9. Who intake more than 14 units of alcohol per week within 3 months prior to screening (1 unit of alcohol= 360 mL of beer, 150 mL of wine or 45 mL of liquor), or have positive result in alcohol breath test (baseline period), or patients who cannot abstain from alcohol during the trial.
10. Who smoke more than 5 cigarettes per day within 3 months prior to screening or have positive results in urine nicotine screening test (screening period or baseline period) or unable to stop using any tobacco products during the trial.
11. Excessive consumption of tea, coffee and/or caffeine-rich beverages (more than 8 cups per day, 1 cup = 250 mL) within 3 months prior to screening.
12. Have participated in another investigational drug trial within 3 months or in 3 or more clinical trials within the last year before the first dose of investigational drug; If the half-life of other investigational drugs is longer, the time interval required will be longer, suggesting 5 half-lives of the investigational drug.
13. Blood donation including blood components or massive blood loss (≥ 200 mL) within 3 months prior to screening; patients who had blood transfusion or have used blood products.
14. Have plan of giving birth or sperm donation within 90 days.
15. Have received vaccine within 4 weeks prior to screening.
16. Have taken any drugs that inhibit or induce hepatic metabolism of the drug within 28 days prior to taking the investigational drug [e.g., barbiturates, carbamazepine, phenytoin, glucocorticoids, omeprazole; SSRI antidepressants, cimetidine, macrolides, nitroimidazoles, sedative hypnotics, fluoroquinolones, antihistamines, antiviral drugs (such as saquinavir, etc.), calcium antagonists (such as diltiazem, verapamil, etc.), rifamycins (such as rifampin, etc.)].
17. Have taken prescription or over-the-counter medicine, dietary supplement or herbal remedy within 14 days prior to the first dose of investigational drug. If the half-life of the concomitant drug is longer, the time interval required will be longer, which is suggested as 5 half-lives of the investigational drug.
18. Any abnormal result in laboratory tests and other examination, which is judged as clinical significance by the investigator.
19. Have positive result in hepatitis B surface antigen, hepatitis B core antibody, hepatitis C antibody, human immunodeficiency virus (HIV) antibody, or Treponema pallidum antibody screening.
20. Have clinically significant abnormality in blood pressure, pulse and body temperature, reference to normal range (including boundary value): blood pressure 90-139/60-89 mmHg; pulse 60-100 bpm; body temperature (ear temperature) 35.4-37.7℃, the specific conditions would be comprehensively determined by the investigator.
21. At screening, corrected QT interval (corrected by Fridericia's formula, QTcF = QT/RR1/3) > 450 msec or QRS complex > 120 msec in 12-lead electrocardiogram (ECG) resting on supine. If QTc exceeds 450 msec or QRS exceeds 120 msec, 2 additional ECG measurements should be repeated, and the subject's eligibility will be determined by using the average value of the 3 QTc or QRS measurements.
22. Unwilling or unable to follow the lifestyle guideline described in the study protocol (e.g. dietary restrictions, activity and contraceptive requirements).
23. Have other acute or chronic medical or psychiatric disease that, in the judgment of the investigator, would make the subject unsuitable or increase the risk associated with participating in this study, or would interfere with interpretation of the study results.
24. Have consumed chocolate, any caffeine-containing, xanthine-containing foods or beverages, and other special diets affecting the absorption, distribution, metabolism, and excretion of the drug during the admission period from screening to Day -2.
25. Inability to keep abstinence from grapefruit or grapefruit-related citrus (e.g. pomelo) fruits or juices within 7 days prior to the first dose of study drug and for the duration of the study.
26. Other subjects, judged by investigators, to be unsuitable for participation in the study.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2019-07-22 (Actual); Primary Completion 2019-09-27 (Actual); Study Completion 2019-09-27 (Actual)

PRIMARY OUTCOMES:
Cmax | 2-month
  Peak Plasma Concentration
Tmax | 2-month
  Time To Reach Maximum Concentration
AUC | 2-month
  Area Under The Curve
t1/2 | 2-month
  Elimination Half-Life

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.03 | 2-month
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.03

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Public Health Clinical Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Meng X, Lin X, Jiang R, Lu Y, Zeng L, Cao M, Zhang J. Effect of Food on the Pharmacokinetics of Senaparib (IMP4297) in Healthy Chinese Subjects. Clin Drug Investig. 2022 Nov;42(11):1009-1016. doi: 10.1007/s40261-022-01198-8. Epub 2022 Oct 14. PMID 36239914